CLINICAL TRIAL: NCT01644162
Title: Use of Ventilator Monitoring for Early Detection of Exacerbations of Chronic Lung Disease
Brief Title: Ventilator Monitoring in Early Exacerbation Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11/LO/1777
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2012-03

CONDITIONS: Respiratory Failure; Neuromuscular Disease; Chest Wall Disorder; Chronic Obstructive Pulmonary Disease; Obesity Hypoventilation Syndrome
Keywords: Non-Invasive Positive-Pressure Ventilation; Disease Exacerbation; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency; Neuromuscular Diseases; Pulmonary Disease, Chronic Obstructive; Obesity Hypoventilation Syndrome; Disease Progression | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iVAPS ventilation (Other): 3 months of ventilator use in iVAPS mode with data monitoring
  Interventions: Device: iVAPS ventilation

INTERVENTIONS:
Device: iVAPS ventilation — 3 months of ventilation on iVAPS mode
  Other Names: non-invasive ventilation

SUMMARY:
The aim of this study is to determine whether respiratory disease exacerbations (a sudden worsening of symptoms) can be predicted by variables that are monitored by non-invasive ventilators (small machines that assist breathing) in patients requiring long term home ventilation.

The investigators hypothesise that acute exacerbations of patients with respiratory disease and ventilatory failure will be predicted by changes in the respiratory variables monitored and stored by ventilators during chronic home ventilator use.

DETAILED DESCRIPTION:
This pilot study is a proof of concept study investigating whether respiratory variables measured during chronic non-invasive ventilation (NIV) therapy may be used to predict a disease exacerbation.

Modern ventilators used in the home for chronic respiratory failure have the ability to monitor and store respiratory variables that may worsen during exacerbations, and may potentially detect exacerbations before symptoms become apparent. Normal pressure support ventilators monitor respiratory rate which might be expected to increase with worsening disease. In patients with obstructive airways disease an increase in expiratory time may potentially be observed with worsening airways obstruction. Adaptive servo ventilators, which modulate pressure support to maintain constant minute ventilation, may increase the amount of pressure support delivered if respiratory mechanics deteriorate as a result of an exacerbation.

Consenting experienced NIV users will be switched to an adaptive-servo ventilator with the capacity to monitor and store therapy data. The device being used is the Stellar 150 ventilator (Resmed, Ltd., Bella Vista, Australia) with hardware and software ability to measure variables such as respiratory rate, airflow, pressure support and leak.

Patients will use the ventilator for a total of 4 months during which they will complete daily symptom diaries, including medication use and peak flow measurements.

Changes in ventilator variables will be analysed and day to day variation identified. Changes will be compared with daily peak expiratory flow measures (an indication of how well the airways are functioning), patient symptoms, and healthcare utilization. Hospital admissions for exacerbations, GP consults, and healthcare team contacts will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of obstructive (COPD, cystic fibrosis, bronchiectasis or chronic asthma) or restrictive (NMD, chest wall disorder) lung disease confirmed by a hospital consultant
* aged > 18 years
* established home ventilator user with ventilator prescribed for either chronic ventilatory failure or nocturnal hypoventilation
* able to use bilevel positive pressure ventilation with Inspiratory positive airway pressure (IPAP) requirement <30cm H2O (Stellar ventilator - IPAP max 30)

Exclusion Criteria:

* patients < 18 years
* cognitive impairment sufficient to interfere with comprehension of the study or use of ventilator
* poor adherence with non-invasive ventilation (<3hours/night for >10days/month)
* Inspiratory positive airway pressure (IPAP) requirement >30cmH2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in ventilator pressure support from baseline | up to 3 months
  Pressure Support delivered by the adaptive-servo ventilator at Day 0 of exacerbation compared to the pressure support during baseline stable state.

SECONDARY OUTCOMES:
Changes in ventilator-measured parameters from baseline | Up to 3 months
  Changes in ventilator-measured parameters >15% from baseline [respiratory rate (RR), inspiratory time (Ti), pressure support (PS), Minute volume (MV), tidal volume (Vt), flow, leak, oxygen saturation (SaO2), pulse, I:E ratio, apnoea-hypopnea index (AHI), compliance]
Exacerbation as determined by a change in patients subjective symptoms | up to 3 months
  The presence of 2 or more subjective symptoms compared to baseline for 2 consecutive days;
  - breathlessness, increased sputum volume or sputum purulence, coryzal, wheeze or chest tightness, sore throat, cough, fever, sleep disruption, decreased physical activity
Change in peak expiratory flow rate (PEFR)>15% from baseline | Up to 3 months
  Change in peak expiratory flow rate (PEFR)>15% from baseline
Exacerbation as defined by healthcare utilisation | up to 3 months
  Exacerbation defined by the requirement of antibiotics +/- steroids, GP visit, accident and emergency visit, hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom